CLINICAL TRIAL: NCT06186882
Title: Gene x Environment Interplay in Developmental Dyslexia Treatment: A Round-trip Translation Between Humans and Animal
Acronym: Gedys
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Università degli studi di Bergamo (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GR-2021-12375102
Record Dates: First submitted 2023-11-30; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Reading Disorder
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ENVIRONMENTAL STIMULATION (Experimental)
  Interventions: Behavioral: Action Video-Game

INTERVENTIONS:
Behavioral: Action Video-Game — Thanks to their specific characteristics (presentation of multiple peripheral, rapidly moving, spatio-temporally unpredictable stimuli), Action Video-Games improve reading skills through their effects on the Magnocellular-Dorsal stream. Training will consist of 20 days of Action Video-Games sessions of 1 hour each, three times per week.

SUMMARY:
Developmental dyslexia affects 7% of school-age children (Male:Female ratio of 1.5:1) and incurs disadvantages in education and occupation. Scientific progress concerning the etiology of developmental dyslexia evidenced the complex gene-environment interaction. The DCDC2-READ1 deletion associates with reading skills and affects the magnocellular-dorsal stream in humans and animals. DCDC2 modifies neural activity within the excitatory pathways. The magnocellular-dorsal stream mediates the function of the attention network. Difficulties in spatial and temporal attention shifting impair letter-to-speech sound integration increasing neural noise. Action video games improve the efficiency of the magnocellular-dorsal stream. The aim of this cutting-edge, round trip translation study is threefold: 1.to unravel new insights behind the pathophysiology of developmental dyslexia, 2. to assess gene-environment interaction effects on developmental dyslexia endophenotypes, and 3. to identify useful clues to foster the identification of new, personalized treatments.

ELIGIBILITY:
Inclusion Criteria

* 5-years old pre-readers,
* normal intelligence quotient,
* no main counter indications for magnetic resonance acquisition,
* no previous diagnosis of any neurodevelopmental disorders.

Exclusion Criteria:

* intelligence quotient below the average range,
* presence of counter indications for magnetic resonance acquisition,
* previous diagnosis of any neurodevelopmental disorders.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Short-term memory | 3 years
  Short-term memory - assessed by the Single Digit Forward Span, Single Digit Backward Span. Measures obtained: Z scores age-corrected.
Phonological awareness | 3 years
  Phonological awareness - assessed by the nonword repetition test. Measures obtained: Z scores age-corrected.
Rapid automatized naming | 3 years
  Rapid automatized naming - assessed by the RAN test. Measures obtained: Z scores age-corrected.
Reading skills | 3 years
  Reading skills - assessed by single unrelated words and pseudo-words reading tests. Measures obtained: Z scores age-corrected.
Visual attention | 3 years
  Visual attention - assessed by a computer-based visual attention task
Visual motion processing | 3 years
  Visual motion processing - assessed by Coherent dot motion task
measurement of neurotransmitters | 3 years
  in vivo measures of neurotransmitters including glutamate and gamma-Aminobutyric acid magnetic resonance spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute IRCCS E Medea, Bosisio Parini, LC, Italy

IPD SHARING:
Plan to Share IPD: No